CLINICAL TRIAL: NCT06710678
Title: Examining Executive Functions in Medical Students Across Different Types of Study Breaks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Amber Sousa, Assistant Professor, New York Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NYIT IRB-2025-152
Record Dates: First submitted 2024-11-21; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Executive Function (Cognition)
Keywords: study breaks; social media; executive function; memory; medical students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Social Media Study Break (Experimental): Medical students will engage in a 10 minute social media study break
  Interventions: Behavioral: Social Media Study Break
- Physical Activity Study Break (Active Comparator): Medical student will engage in a 10 minute light physical activity study break
  Interventions: Behavioral: Physical Activity Study Break
- No study break (No Intervention): Medical students will continue to study instead of a break

INTERVENTIONS:
Behavioral: Physical Activity Study Break — A 10-minute walking/upper extremity light movement indoor break from study session
  Arms: Physical Activity Study Break
Behavioral: Social Media Study Break — Participants will engage in social media use/engagement during a 10-minute study session break
  Arms: Social Media Study Break

SUMMARY:
This study aims to expand on previous findings and compare the effects of an active break (ten minutes of walking or upper body movement), a digital break (ten minutes of phone use), and no break on memory and attention in medical students after a prolonged period of studying. The List Learning Task, Stroop Test, and Sustained Attention to Response Task will be administered to measure memory, executive function, and attention, respectively. Information on how different types of breaks affect memory and attention may prompt medical students to be more mindful and intentional of the way they spend their time in between studying.

DETAILED DESCRIPTION:
120 people will be recruited. Following consent procedures, those who choose to participate will be randomized to physical intervention, digital intervention or control. 40 will be randomly selected to be in the active physical break group, another 40 participants will selected to be in the passive digital break group, and another 40 will be selected to be in the group without any break.

All participants will complete a demographic form and a baseline Stroop and Sustained Attention to Response Task tests prior to starting the experiment. Next, participants in all three groups will self-study any form of class material for 45 minutes without any breaks or phone usage. At the 45 min mark, the first part of the List Learning Task will be administered to all participants. Following completion, participants in the active physical break and passive digital break groups will begin their 15 min breaks. Those in the former group will engage in 10 min of walking or upper body movement. Those in the latter group will engage in 10 min of social media usage. An additional 5 min will be allotted to allow participants to get settled after their break and use the bathroom if needed before continuing with the study. Participants in the control group will continue studying for 15 min. All participants will not be permitted to converse or interact with each other throughout the break. Once the 15 min break has concluded, all participants will be administered the second part of the List Learning Task. When that is completed, participants will be given the Stroop Test and Sustained Attention to Response Task. A survey will be given to the passive digital break group to determine which social media app(s) were used. All groups will be surveyed about their thoughts regarding their respective type of break or lack thereof and its effect on their studying.

ELIGIBILITY:
Inclusion Criteria:

* have and regularly use some form of social media
* able to perform light physical activity such as walking or upper body movement

Exclusion Criteria:

* no social media usage
* color blindness (cognitive tests require color perception)
* ADHD or other known conditions that affect attention and/or concentration,
* current concussion
* any condition that prevents upper or lower body physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Sustained Attention to Response Task | from enrollment until the end of their partipation which lasts one day
  Sustained Attention to Response Task is a go/nogo task with infrequent nogo signals to measure attention. Participants are presented with a single digit 1-9 in the middle of the screen in varying font sizes. The digit disappears after a short while and is replaced with a mask (circle with an X). Participants are asked to press the SPACEBAR if any digit other than 3 is presented and to withhold the response if digit 3 is presented.

SECONDARY OUTCOMES:
Stroop Task | from enrollment until the end of their partipation which lasts one day
  The classic Stroop paradigm demonstrates the interference of word meaning on the naming of the color in which the words are written as measured by reaction time/accuracy differences to color-meaning congruent and color-meaning incongruent combinations. Participants are given color words written in color and are asked to indicate the color of the word (not its meaning) by key press as fast as they can without making too many errors. Congruent trials: color word and the color it is presented in are the same Incongruent trials: color word and the color it is presented in are not the same Control trials: colored rectangles.
List Learning Task | from enrollment until the end of their partipation which lasts one day
  The List Learning Task is a basic computer-adapted List Learning Task inspired by the one used by The Repeatable Battery for Neuropsychological Status (RBANS). The script presents the list visually and accepts written input.
  Participants are presented a list of words (fixed sequence), one at a time, on the computer screen. Once the list has finished, a textbox appears and participants are asked to enter as many of the list words as they remember, in any order. The list learning/recall task is repeated 3 more times before a break (default: 15min). After the break, participants work through an optional delayed recall test and a recognition task: 20 words are presented to them, one by one, and participants have to decide whether the word was part of the orinal list.

CONTACTS AND LOCATIONS:
Overall Officials: Amber Sousa, PhD, Principal Investigator — NYIT COM
Locations (1):
- NYIT, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No